CLINICAL TRIAL: NCT06646588
Title: Fruquintinib in Combination With Tislelizumab Followed by Radiotherapy in Relapsed or Progressive Esophageal Squamous Cell Carcinoma
Brief Title: Fruquintinib in Combination With Tislelizumab Followed by Radiotherapy in Esophageal Squamous Cell Carcinoma
Acronym: SJZ-RMEEC01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJZ-RMEEC01
Record Dates: First submitted 2024-10-07; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Neoplasms
MeSH Terms: conditions — Esophageal Neoplasms | interventions — HMPL-013; tislelizumab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib in Combination With Tislelizumab followed by radiotherapy (Experimental): Fruquintinib in Combination With Tislelizumab followed by radiotherapyin Relapsed or Progressive Esophageal Squamous Cell Carcinoma
  Interventions: Drug: Fruquintinib; Drug: Tislelizumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib: Oral, once daily, 2 weeks on and 1 week off. The product can be taken with food or orally on an empty stomach, and needs to be swallowed whole. It is recommended that the dose be taken at the same time each day; if the patient vomits after taking the dose, no refill is needed; a missed dose should not be added the next day, but the next prescribed dose should be taken as usual.
Drug: Tislelizumab — Tislelizumab: intravenous drip 200mg，day1，once every three weeks.
Radiation: Radiotherapy — Radiotherapy synchronised with drugs.

SUMMARY:
According to the Global Burden of Disease Study, the number of esophageal cancer cases globally increased from 319,969 in 1990 to 534,563 in 2019, a relative increase of 67.07 per cent. In addition, GLOBOCAN 2020 reported that the global incidence of esophageal cancer climbed to 604,100, accounting for 3.1% of all tumor sites and ranking 7th out of 36 cancers. In addition, the number of global deaths from esophageal cancer increased from 319,332 in 1990 to 498,067 in 2019, a relative increase of 55.97%.GLOBOCAN 2020 reported about 544,076 new esophageal cancer deaths, which accounted for 5.5% of all study centres and ranked 6th among 36 cancers. Chemotherapy is the standard of care for advanced esophageal squamous cell carcinoma, but conventional chemotherapy has limited efficacy, and studies have shown lower median overall survival with chemotherapy in patients with advanced esophageal cancer compared to patients with other stages. In recent years, with the first-line approval of immune checkpoint inhibitors, the treatment of esophageal cancer has entered the immune era. Immune checkpoint inhibitors have become an important therapeutic option for patients with advanced esophageal cancer who have failed chemotherapy. This study will explore the efficacy and safety of this small molecule anti-angiogenic drug, fruquintinib, in combination with tislelizumab in esophageal squamous cell carcinoma previously treated with immune checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and written signed informed consent;
* Age ≥ 18 years old, gender is not limited;
* Histologically or cytologically confirmed limited-stage small cell lung cancer (2009 AJCC/UICC/IASLC lung cancer TNM staging criteria, limited-stage SCLC is any T stage, any N stage, and M0), and patients with suspected brain or bone metastasis at the time of screening should undergo brain MRI or ECT before study enrollment;
* There are immunohistochemical results;
* Chemotherapy must include either cisplatin or carboplatin, in combination with etoposide;
* Physical status score ECOG 0-1;
* Weight > 40 kg;
* Expected survival ≥ 6 months;
* According to RECIST 1.1 guidelines, at least one lesion (not previously receiving radiotherapy) with a maximum diameter ≥ 10 mm as accurately measured by computed tomography (CT) or magnetic resonance imaging (MRI) at baseline (except lymph nodes, whose short axis must be ≥ 15 mm); And the lesion is suitable for repeated accurate measurement.;
* No previous immunotherapy;
* no serious abnormalities of haematopoietic, cardiac, pulmonary, hepatic; and renal functions and immunodeficiency (Haematology: white blood cells ≥3.5×109/L; neutrophils ≥1.5×109/L; haemoglobin ≥90g/L; platelets

  ≥100×109/L. Liver and kidney function: total bilirubin ≤1.5 times the upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) ≤2.5 times the upper limit of normal; creatinine ≤1.5 times the upper limit of normal; albumin ≥30 g/L. Coagulation: International Normalised Ratio (INR) or Prothrombin Time (PT) or Activated Partial Thromboplastin Time (APTT)

  ≤ 1.5 times ULN; if the subject is receiving anticoagulation therapy, PT or INR is acceptable as long as the PT or INR is within the range of the anticoagulant drug formulation. Echocardiographic assessment: left ventricular ejection fraction (LVEF) ≥ low limit of normal (50%). Pulmonary function FEV1 ≥70% of % of predicted value and DLCO ≥60% of % of predicted value).
* The female patient has evidence of postmenopausal status, or the urine or serum pregnancy test results of the premenopausal woman are negative. Women who stop menstruating for 12 months without other medical reasons are considered menopausal.

Exclusion Criteria:

* Distant organ metastases (excluding supraclavicular lymph nodes) as determined by CT evaluation during screening and prior imaging;
* have received prior radiotherapy to the chest;
* have medical contraindications to etoposide - platinum (carboplatin or cisplatin) based chemotherapy;
* having any active autoimmune disease or a history of autoimmune disease (e.g. interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (which can be included if hormone replacement therapy is effective), etc.), and a history of immunosuppressive drug use within 28 days, with the exception of the use of hormones for the purpose of dealing with toxicity from radiotherapy;
* Previously received or are receiving other PD-1 antibody therapy or other immunotherapy targeting PD-1/PD-L1, or are currently participating in other interventional clinical studies for treatment;
* Have received other anti-tumour therapy (including herbal therapy with anti-tumour effect) within 4 weeks prior to the first dose of the study; have received long-term systemic immunotherapy or hormone therapy (except physiological replacement therapy, e.g., oral thyroxine for hypothyroidism) within 4 weeks prior to the first dose of the study; and have been treated with other experimental drugs or interventional clinical studies within 4 weeks prior to the first dose of the study;
* Patients with uncontrolled clinical cardiac symptoms or disease such as

  (1) NYHA class II or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, and (4) clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
* with congenital or acquired immune function defects (e.g., HIV-infected patients), active hepatitis B (HBV-DNA ≥104 copies/ml) or hepatitis C (hepatitis C antibody-positive with HCV-RNA above the lower limit of detection of the analytical method), or active tuberculosis;
* Have an active infection or unexplained fever >38.5°C within 2 weeks prior to screening (at the investigator's discretion, subjects may be enrolled for fever arising from tumours);
* In the judgement of the investigator, the subject has other factors that may cause him/her to be forced to terminate the study in the middle of the study, e.g., suffering from other serious illnesses (including psychiatric illnesses) that require comorbid treatment, family or social factors that may affect the safety of the subject or the collection of trial data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of objective remission rate (ORR) in Relapsed or Progressive Esophageal Squamous Cell Carcinoma patients receiving Fruquintinib in Combination With Tislelizumab Followed by Radiotherapy | at least 2 years
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). Objective remission rate (ORR): defined as the proportion of subjects whose tumor volume shrinks to a pre-specified value and can be maintained for the minimum time frame required, incorporating cases in complete remission (CR) and partial remission (PR).

SECONDARY OUTCOMES:
Assessment of disease control rate (DCR) in Relapsed or Progressive Esophageal Squamous Cell Carcinoma patients receiving Fruquintinib in Combination With Tislelizumab Followed by Radiotherapy | at least 2 years
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). Disease control rate (DCR): the proportion of patients whose tumors shrank or were stable and remained so for a certain period of time, including complete remission (CR), partial remission (PR) and stable disease (SD).
Assessment of overall survival (OS) in Relapsed or Progressive Esophageal Squamous Cell Carcinoma patients receiving Fruquintinib in Combination With Tislelizumab Followed by Radiotherapy | at least 2 years
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). OS is defined as the time from the start of enrollment to death from any cause.
Assessment of progression-free survival (PFS) in Relapsed or Progressive Esophageal Squamous Cell Carcinoma patients receiving Fruquintinib in Combination With Tislelizumab Followed by Radiotherapy | at least 2 years
  Objective tumor remission is assessed by the investigator using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria). PFS is defined as the time from the start of enrollment until tumor progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China